CLINICAL TRIAL: NCT03248882
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING, PARALLEL GROUP STUDY TO EVALUATE SAFETY, TOLERABILITY, AND PHARMACODYNAMICS OF PF-05221304 ADMINISTERED DAILY FOR 16-WEEKS TO ADULT SUBJECTS WITH NONALCOHOLIC FATTY LIVER DISEASE
Brief Title: Phase 2a, Dose-ranging Study With PF-05221304 in Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C1171002; 2017-001156-55 (EudraCT Number)
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Results first posted 2020-03-10 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-02

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
Keywords: PF-05221304; NAFLD; NASH; features of metabolic syndrome; Dose-Ranging Study
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: C1171002 is a randomized, double blind, placebo controlled, 5 arm (placebo, plus 4 active doses of PF 05221304), parallel group study.
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Double-Blind, PF-05221304-matching Placebo
  Interventions: Drug: Placebo
- PF-05221304 - 2 mg (Active Comparator): PF-05221304 - 2 mg, once-daily
  Interventions: Drug: PF-05221304
- PF-05221304 - 10 mg (Active Comparator): PF-05221304 - 10 mg, once-daily
  Interventions: Drug: PF-05221304
- PF-05221304 - 25 mg (Active Comparator): PF-05221304 - 25 mg, once-daily
  Interventions: Drug: PF-05221304
- PF-05221304 - 50 mg (Active Comparator): PF-05221304 - 50 mg, once-daily
  Interventions: Drug: PF-05221304

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-05221304 — PF-05221304, Experimental Drug
  Arms: PF-05221304 - 10 mg; PF-05221304 - 2 mg; PF-05221304 - 25 mg; PF-05221304 - 50 mg

SUMMARY:
Phase 2a, dose-ranging Study with PF-05221304 in Nonalcoholic Fatty Liver Disease (NAFLD)

DETAILED DESCRIPTION:
A Phase 2a, Randomized, Double-blind, Placebo-controlled, Dose-ranging, Parallel Group Study To Evaluate Safety, Tolerability, And Pharmacodynamics Of PF-05221304 Administered Daily For 16-weeks To Adult Subjects With Nonalcoholic Fatty Liver Disease

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >= 25 kg/m2
* Body Weight > 50 kg
* Liver fat (assessed via MRI-PDFF) >= 8%
* Biopsy-proven NASH - diagnosed in previous 24-months
* Presumed NASH - per Sponsor's definition
* NAFLD with minimal inflammation/fibrosis
* Features of Metabolic Syndrome

Exclusion Criteria:

* Alcohol-induced steatohepatitis or other forms of chronic liver disease
* Positive for Hepatitis B, Hepatitis C, or Human Deficiency Virus
* Severe Renal Impairment
* Contraindications for MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (138):
- United States (60):
  - Franco Felizarta MD, Bakersfield, California
  - eStudySite, Chula Vista, California
  - San Diego Imaging Chula Vista, Chula Vista, California
  - University of California, San Diego (Altman Clinical and Translational Research Institute), La Jolla, California
  - University of California, San Diego, La Jolla, California
  - eStudySite, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - National Research Institute, Los Angeles, California
  - Stanford University Medical Center, Blake wilbur Building, Palo Alto, California
  - Stanford University Medical Center, Palo Alto, California
  - Huntington Medical Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - Precision Research Institute, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - South Denver Gastroenterology, P.C., Englewood, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Stand Up MRI of Miami, Miami, Florida
  - Ocean Blue Medical Research Center, Inc, Miami Springs, Florida
  - Avail Clinical Research, LLC, Orange City, Florida
  - Bioclinica Research, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Tampa General Medical Group, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - South Florida Center Of Gastroenterology, PA, Wellington, Florida
  - Independent Imaging, Wellington, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Invision Imaging, Honolulu, Hawaii
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Ascension Via Christi Imaging at St. Francis, Wichita, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic- Main Campus, Rochester, Minnesota
  - Gastrointestinal Associates, PA, Flowood, Mississippi
  - Colonnades at Baptist, Jackson, Mississippi
  - BioTelemetry Research, Rochester, New York
  - Investigational Drug Service, University of North Carolina Hospitals, Chapel Hill, North Carolina
  - The University of NC at Chapel Hill, Clinical and Translational Research Center (CTRC), Chapel Hill, North Carolina
  - The University of North Carolina at Chapel Hill, Biomedical Research Imaging Center (MRI Facility), Chapel Hill, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research, Inc., Winston-Salem, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Prime Imaging (Chattanooga Outpatient Center), Chattanooga, Tennessee
  - ClinSearch, Chattanooga, Tennessee
  - Touchstone, Austin, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Pinnacle Clinical Research, Rollingwood, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Pinnacle Clinical Research, PLLC, San Antonio, Texas
  - Clinical Research Advantage, Inc./Wasatch Peak Family Practice, Layton, Utah
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
- Australia (9):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Spectrum Medical Imaging, Randwick, New South Wales
  - Castlereagh Imaging, Westmead, New South Wales
  - Storr Liver Centre, Westmead Hospital, Westmead, New South Wales
  - Dr. Jones & Partners Medical Imaging, Adelaide, South Australia
  - Royal Adelaide Hospital, Department of Gastroenterology and Hepatology, Adelaide, South Australia
  - Flinders Medical Centre/Department of Gastroenterology & Hepatology, Adelaide, South Australia
  - Radiology SA, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (38):
  - Dr TG Elliott Inc - BC Diabetes, Vancouver, British Columbia
  - False Creek Healthcare Centre, Vancouver, British Columbia
  - False Creek Healthcare, Vancouver, British Columbia
  - LAIR Centre, Vancouver, British Columbia
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - West Coast Medical Imaging, Victoria, British Columbia
  - Nova Scotia Health Authority, QEII Health Sciences Centre, Halifax, Nova Scotia
  - Nova Scotia Health Authority - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - St. Joseph's Health Care London, London, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Oxford Medical Imaging, Mississauga, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - St. Michael's Hospital - MRI Research Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network (UHN) - Toronto General Hospital - Toronto Centre for Liver Disease (TCLD), Toronto, Ontario
  - University of Toronto - Toronto General Hospital, Toronto, Ontario
  - University Health Network (UHN), Toronto, Ontario
  - Toronto Liver Centre - Liver Care Centre Corporation, Toronto, Ontario
  - Resonance Magnetique du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Medpharmgene Inc, Montreal, Quebec
  - Clinique de Medecine Urbaine du Quartier Latin, Montreal, Quebec
  - Centre de recherche du CHUM, Montreal, Quebec
  - Cedar Cancer Center - McGill University Health Centre, Montreal, Quebec
  - Chronic Viral Illness Service - Royal Victoria Hospital - McGill University Health Centre (MUHC), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Research Institute of the MUHC, Montreal, Quebec
  - Radiologie Varad, Montreal, Quebec
  - IRM Quebec, Québec, Quebec
  - CHU de Quebec - Universite Laval - site Centre Hospitalier de l'Universite Laval (CHUL), Québec, Quebec
  - Centre de recherche de l'Institut Universitaire de Cardiologie et de pneumologie de Quebec, Québec, Quebec
  - Centre de recherche Saint-Louis, Québec, Quebec
  - IRM Québec - Clinique St-Louis, Québec, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - Clinix, Québec, Quebec
  - Recherche Medicale St-Jerome Inc, Saint-Jérôme, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux (CIUSSS) de l'Estrie, Sherbrooke, Quebec
- Israel (10):
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Hebrew University Medical Center - Ein Kerem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Poland (16):
  - ClinicMed Badurski i wspolnicy Spolka Jawna, Bialystok
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Osrodek Badan Klinicznych, Jaworze
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Silmedic Sp. z o.o. Oddzial w Katowicach, Katowice
  - Centrum Medyczne A-Z Clinic, Krakow
  - Krakowskie Centrum Medyczne sp. z o.o., Krakow
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Synexus Polska Sp. z o.o Oddzial w Poznaniu, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Synexus Polska Sp. z o. o. Oddzial w Warszawie, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Badan Klinicznych, Wroclaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - DOBROSTAN - Gabinety Lekarskie, Wroclaw
- Taiwan (5):
  - Changhua Christian Hospital, Changhua, Changhua County
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sivakumar P, Saul M, Robinson D, King LE, Amin NB. SomaLogic proteomics reveals new biomarkers and provides mechanistic, clinical insights into Acetyl coA Carboxylase (ACC) inhibition in Non-alcoholic Steatohepatitis (NASH). Sci Rep. 2024 Jul 24;14(1):17072. doi: 10.1038/s41598-024-67843-8. PMID 39048608
- [Derived] Calle RA, Amin NB, Carvajal-Gonzalez S, Ross TT, Bergman A, Aggarwal S, Crowley C, Rinaldi A, Mancuso J, Aggarwal N, Somayaji V, Inglot M, Tuthill TA, Kou K, Boucher M, Tesz G, Dullea R, Bence KK, Kim AM, Pfefferkorn JA, Esler WP. ACC inhibitor alone or co-administered with a DGAT2 inhibitor in patients with non-alcoholic fatty liver disease: two parallel, placebo-controlled, randomized phase 2a trials. Nat Med. 2021 Oct;27(10):1836-1848. doi: 10.1038/s41591-021-01489-1. Epub 2021 Oct 11. PMID 34635855
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1171002

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to PF-05221304 tablet was administered orally once daily (QD) for up to 16 weeks.
- PF-05221304 2 mg: PF-05221304 tablet was administered orally at 2 mg QD for up to 16 weeks.
- PF-05221304 10 mg: PF-05221304 tablet was administered orally at 10 mg QD for up to 16 weeks.
- PF-05221304 25 mg: PF-05221304 tablet was administered orally at 25 mg QD for up to 16 weeks.
- PF-05221304 50 mg: PF-05221304 tablet was administered orally at 50 mg QD for up to 16 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
Started | 61 | 63 | 62 | 58 | 61
Received Treatment | 61 | 63 | 62 | 58 | 61
Completed | 54 | 58 | 55 | 48 | 48
Not Completed | 7 | 5 | 7 | 10 | 13
Not completed — Adverse Event | 3 | 3 | 2 | 6 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of randomized study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg | Total
Number analyzed (Participants) | 61 | 63 | 62 | 58 | 61 | 305
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (10.8) | 54.1 (11.9) | 52.7 (12.8) | 54.0 (11.6) | 52.8 (13.1) | 53.38 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 33 | 35 | 30 | 171
  Male | 25 | 26 | 29 | 23 | 31 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 53 | 50 | 52 | 46 | 51 | 252
  Black or African American | 1 | 1 | 1 | 1 | 0 | 4
  Asian | 5 | 7 | 7 | 9 | 10 | 38
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  Not Reported | 2 | 3 | 2 | 2 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Liver Fat by Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI- PDFF) at Week 16
Description: MRI-PDFF utilized a gradient echo sequence with low flip angle (FA) to minimize T1 bias, corrected T2* decay (due to iron overload) via modeling of the fat signal as a superposition of multiple frequency components from 5 different lipid types, and was applied in each of the 9 Couinaud segments. This technique improved fat quantification accuracy for the entire liver permitting quantification of small differences/changes following pharmacological intervention.
Time Frame: Baseline (between Day -14 and Day 1), Week 16
Population: All randomized participants who received at least 1 dose of randomized study treatment and with non-missing baseline and post-baseline endpoint.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
Number analyzed (Participants) | 55 | 59 | 57 | 54 | 51
Percent change | -7.2 [-13.9 to 0.0] | -17.1 [-22.7 to -11.1] | -49.9 [-53.3 to -46.2] | -55.9 [-59.0 to -52.4] | -64.8 [-67.5 to -62.0]
Statistical Analysis 1: Comparison: Placebo vs PF-05221304 2 mg; Test type: Superiority; Mean Difference (Net) = -10.7, 80% CI 2-sided [-19.4 to -1.1]
Statistical Analysis 2: Comparison: Placebo vs PF-05221304 10 mg; Test type: Superiority; Mean Difference (Net) = -46.0, 80% CI 2-sided [-51.3 to -40.1]
Statistical Analysis 3: Comparison: Placebo vs PF-05221304 25 mg; Test type: Superiority; Mean Difference (Net) = -52.4, 80% CI 2-sided [-57.2 to -47.1]
Statistical Analysis 4: Comparison: Placebo vs PF-05221304 50 mg; Test type: Superiority; Mean Difference (Net) = -62.1, 80% CI 2-sided [-66.0 to -57.8]

2. Secondary Outcome: Percent Change From Baseline in Alanine Aminotransferase at Week 16
Description: Potential improvement in liver function was denoted by reduction in alanine transaminase (ALT)
Time Frame: Baseline (Day 1 pre-dose), Week 16
Population: All randomized participants who received at least 1 dose of randomized study treatment and diagnosed/presumed with nonalcoholic steatohepatitis.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
Number analyzed (Participants) | 40 | 42 | 42 | 39 | 40
Percent change | -8.5 [-15.2 to -1.2] | -12.5 [-18.7 to -5.8] | -27.7 [-32.9 to -22.2] | -31.3 [-36.6 to -25.5] | -46.8 [-50.8 to -42.4]
Statistical Analysis 1: Comparison: Placebo vs PF-05221304 2 mg; Test type: Superiority; Mean Difference (Net) = -4.4, 80% CI 2-sided [-14.0 to 6.3]
Statistical Analysis 2: Comparison: Placebo vs PF-05221304 10 mg; Test type: Superiority; Mean Difference (Net) = -21.0, 80% CI 2-sided [-29.0 to -12.2]
Statistical Analysis 3: Comparison: Placebo vs PF-05221304 25 mg; Test type: Superiority; Mean Difference (Net) = -25.0, 80% CI 2-sided [-32.8 to -16.1]
Statistical Analysis 4: Comparison: Placebo vs PF-05221304 50 mg; Test type: Superiority; Mean Difference (Net) = -41.8, 80% CI 2-sided [-47.9 to -35.0]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a study subject administered a product or medical device. A serious AE (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Any such events with initial onset or increasing in severity after the first dose of study treatment were counted as treatment-emergent.
Time Frame: From first dose of study treatment (Day 1) up to Week 20
Population: All randomized participants who received at least 1 dose of randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
Number analyzed (Participants) | 61 | 63 | 62 | 58 | 61
Participants
  All-causality AE | 41 | 40 | 42 | 45 | 40
  All-causality SAE | 0 | 1 | 1 | 2 | 2
  Treatment-related AE | 16 | 9 | 12 | 16 | 23
  Treatment-related SAE | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology (hemoglobin, hematocrit, erythrocytes, reticulocytes, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes, activated partial thromboplastin time, prothrombin time [PT], PT/international normalized ratio, reticulocytes); chemistry (indirect bilirubin, direct bilirubin, protein, albumin, blood urea nitrogen, creatinine, creatine kinase, urate, calcium, sodium, potassium, chloride, bicarbonate, urine urobilinogen); urinalysis (pH, urine glucose, urine ketones, urine protein, urine hemoglobin, nitrites, leukocyte esterase, urine erythrocytes, urine leukocytes, urine hyaline casts, urine bilirubin, granular casts).
Time Frame: From first dose of study treatment (Day 1) up to Week 20
Population: All randomized participants who received at least 1 dose of randomized study treatment and had laboratory data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
Number analyzed (Participants) | 59 | 63 | 62 | 58 | 61
Participants | 39 | 44 | 36 | 33 | 40

5. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Predefined Criteria
Description: Vital signs categorical summarization criteria: 1) sitting systolic blood pressure (SBP) <90 or >180 millimeters of mercury (mmHg); 2) sitting diastolic blood pressure (DBP) <50 mmHg or >110 mmHg; 3) sitting pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in sitting DBP greater than or equal to (>=) 20 mmHg; 5) change from baseline (increase or decrease) in sitting SBP >=30 mmHg.
Time Frame: From first dose of study treatment (Day 1) up to Week 18
Population: All randomized participants who received at least 1 dose of randomized study treatment and had vital signs data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
Number analyzed (Participants) | 60 | 63 | 62 | 58 | 61
Participants
  Sitting SBP <90 mmHg | 0 | 0 | 0 | 0 | 2
  Sitting SBP >180 mmHg | 0 | 0 | 0 | 1 | 0
  Sitting SBP increase >=30 mmHg | 5 | 6 | 2 | 2 | 0
  Sitting SBP decrease >=30 mmHg | 2 | 1 | 5 | 7 | 6
  Sitting DBP <50 mmHg | 1 | 0 | 0 | 0 | 0
  Sitting DBP >110 mmHg | 0 | 0 | 0 | 0 | 1
  Sitting DBP increase >=20 mmHg | 1 | 4 | 2 | 2 | 3
  Sitting DBP decrease >=20 mmHg | 0 | 4 | 3 | 4 | 4
  Sitting pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0
  Sitting pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With 12-Lead Electrocardiogram (ECG) Data Meeting Predefined Criteria
Description: ECG categorical summarization criteria: 1) QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization) >=140 milliseconds (msec); 2) QRS interval >=50% change from baseline; 3) PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization) >=300 msec; 4) PR interval >=25% change when baseline is >200 msec or >=50% change when baseline is <=200 msec; 5) QT interval (time from ECG Q wave to the end of the T wave corresponding to electrical systole): absolute value of >=500 msec; 6) QTcF interval (QT corrected for heart rate using Fridericia's formula) absolute value of 450 to <480 msec; 7) QTcF interval: absolute value of 480 to <500 msec; 8) QTcF interval: absolute value >=500 msec; 9) QTcF interval: a change from baseline of 30 to <60 msec; 10) QTcF interval: a change from baseline >=60 msec.
Time Frame: From first dose of study treatment (Day 1) up to Week 18
Population: All randomized participants who received at least 1 dose of randomized study treatment and had ECG data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
Number analyzed (Participants) | 60 | 63 | 61 | 58 | 60
Participants
  PR interval >=300 msec | 0 | 0 | 0 | 0 | 0
  %Change in PR interval >=25/50% | 0 | 1 | 0 | 1 | 1
  QRS interval >=140 msec | 0 | 0 | 1 | 0 | 0
  %Change in QRS interval >=50% | 0 | 0 | 0 | 0 | 0
  QT interval >=500 msec | 0 | 0 | 0 | 1 | 0
  QTcF interval >=450 to <480 msec | 6 | 10 | 7 | 9 | 3
  QTcF interval >=480 to <500 msec | 0 | 1 | 0 | 1 | 1
  QTcF interval >=500 msec | 0 | 0 | 0 | 0 | 0
  QTcF interval increase >=30 to 60 msec | 5 | 6 | 8 | 10 | 4
  QTcF interval increase >=60 msec | 2 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 20 weeks
Arm/Group | Placebo | PF-05221304 2 mg | PF-05221304 10 mg | PF-05221304 25 mg | PF-05221304 50 mg
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/63 | 0/62 | 0/58 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/63 | 1/62 | 2/58 | 2/61
Other Adverse Events (participants affected / at risk) | 27/61 | 21/63 | 25/62 | 31/58 | 29/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | PF-05221304 2 mg (N=63) | PF-05221304 10 mg (N=62) | PF-05221304 25 mg (N=58) | PF-05221304 50 mg (N=61)
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | PF-05221304 2 mg (N=63) | PF-05221304 10 mg (N=62) | PF-05221304 25 mg (N=58) | PF-05221304 50 mg (N=61)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 8 | 2 | 4
Nausea (Gastrointestinal disorders) | 3 | 0 | 3 | 5 | 4
Fatigue (General disorders) | 5 | 3 | 2 | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 3 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 3 | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 5 | 4
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 3 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1 | 6 | 4 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 2 | 1
Dizziness (Nervous system disorders) | 4 | 3 | 1 | 3 | 3
Headache (Nervous system disorders) | 8 | 3 | 3 | 7 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT03248882/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03248882/SAP_001.pdf